CLINICAL TRIAL: NCT07198048
Title: Treating Attention and Language in Post-stroke Aphasia Using a Music-based Intervention.
Brief Title: Can Listening to Music Improve Attention and Language After Post-Stroke Aphasia?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, LaCroixLab, Assistant Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-1005; 25PTA147785 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Aphasia; Stroke; Stroke and Aphasia; Stroke Hemorrhagic; Stroke Ischemic; Music Intervention
Keywords: stroke; aphasia; attention; language; music; music intervention
MeSH Terms: conditions — Aphasia; Stroke; Hemorrhagic Stroke; Ischemic Stroke; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Based Intervention (Experimental): Participants in this arm will participate in the music intervention. For this intervention, participants will work with a music therapist and attend to music for 30 minutes each day over the course of 10 weeks.
  Interventions: Behavioral: Music-Based Therapy for Post Stroke Aphasia
- Audiobook listeners (Active Comparator): Participants in this arm will participate in the audiobook intervention. For this intervention, participants will work with a speech-language pathologist and attend to audiobooks for 30 minutes each day over the course of 10 weeks.
  Interventions: Behavioral: Audiobook Intervention for Post Stroke Aphasia
- No Contact Control (No Intervention): The no-contact control arm is designed to demonstrate that any behavioral changes observed in the experimental (MBI) arm are due to the intervention itself, rather than spontaneous recovery processes. While PWA did not achieve full recovery through spontaneous processes, they may still experience improvements over time that occur independently of therapeutic interventions. The use of a no-contact control arm allows us to determine whether any changes observed in the experimental arm exceed those that might naturally occur without participation in the intervention.

INTERVENTIONS:
Behavioral: Music-Based Therapy for Post Stroke Aphasia — Participants will be instructed to maintain their usual activities each day, except we will ask them to select a time of day, a comfortable and distraction free environment, and an apparatus for regular music listening (earbuds, headphones, speakers). Participants will listen mindfully to randomized selections from the playlist that meets their needs that day (i.e., energizing or relaxing). Participants will listen to their music selections on shuffle for 30 minutes per day for 8 weeks using the strategies provided by the music therapist. The target listening duration is 30 minutes as it is a common target for time spent on task before taking a break. Participants will complete their daily journal entry immediately after music listening. The music therapist will make a weekly telephone call to each participant in the experimental arm. The telephone call will last ~30 minutes. During this telephone call, the music therapist will update the music playlists and help submit their logs.
  Arms: Music Based Intervention
Behavioral: Audiobook Intervention for Post Stroke Aphasia — Participants will be instructed to maintain their usual activities each day, except we will ask them to select a time of day, a comfortable and distraction free environment, and an apparatus for regular music listening (earbuds, headphones, speakers). Participants will listen mindfully to an audiobook selected with a speech-language pathologist (SLP). Participants will listen to their audiobook for 30 minutes per day for 8 weeks using the strategies provided by the SLP. The target listening duration is 30 minutes as it is a common target for time spent on task before taking a break. Participants will complete their daily journal entry immediately after audiobook listening. The SLP will make a weekly telephone call to each participant in the experimental arm. The telephone call will last ~30 minutes. During this telephone call, the SLP will update the audiobook library and help submit their logs.
  Other Names: Active Control
  Arms: Audiobook listeners

SUMMARY:
The goal of this clinical trial is to learn if a music-based intervention can acutely improve three types of attention (alerting, orientating, executive control) in people with aphasia following a stroke.

The main questions it aims to answer are:

1. Is a music based intervention effective at improving attention with someone who has aphasia?
2. Does music-induced changes in attention improve language abilities and quality of life with someone who has aphasia? Researchers will compare a group that listening to music, to listing to an audiobook group, to a group that serves as a control to see if there are changes in attention over time.

Participants will:

1. Listen to music or an audiobook for 30 minutes a day for 8 weeks
2. Complete a daily journal about each day's listening experience
3. Complete three testing sessions where attention, language, and quality of life are assessed.

DETAILED DESCRIPTION:
Participants: Participants will be 45 people with aphasia (PWA) who are a representative sample of the diversity of the Lafayette, Indiana area, and broader United States. We will recruit PWA from the PI's research registry, which includes ~60 PWA, Purdue's in-house Speech, Language, and Hearing clinics, local assisted living and rehabilitation hospitals, public community centers, and online. The PI has extensive experience recruiting from these sources and recently recruited 43 PWA for a similar study in one year. PWA will be included in the study if they are 18+ years of age, had a stroke at least 6 months prior to study enrollment, have normal or corrected to normal hearing and vision, no history of an attention disorder pre-stroke, and at least a mild aphasia on the Western Aphasia Battery Revised (WAB-R). Hearing acuity will be screened using pure tone audiometry at 500-4000 Hz. Vision will be assessed using self assessment Randomization to Study Arms: Participants will be randomly assigned to either the experimental arm, active control arm, or the no-contact control arm (n = 15 per arm). The study arms are adapted from a previous study in which acute stroke survivors listened to music, an audiobook, or no prescribed auditory material daily over an 8-week period. However, PWA are a distinct clinical population from acute stroke warranting a specific investigation into whether the MBI similarly impacts attention in PWA, and subsequently their language abilities and quality of life.

Experimental Arm: Receptive Music-Based Intervention In an initial one-hour meeting, a board-certified music therapist will work with each participant to assess their music preferences and curate two playlists using the Spotify Music app. One playlist will include highly energizing pieces. The second playlist will include relaxing pieces. The playlists will include music selected by the participant and music by the same or similar artists, instrumentation, or genres, and will be chosen in consultation with the music therapist. The lists will be of sufficient length to allow the selections to be shuffled for listening each day without repetition based on the previous day's listening.

In a second one-hour meeting, the music therapist will teach the participant listening techniques to help them attend closely to the music and observe its effects on their mind and body, including movements, associations, memories, images, breathing rate, and levels of relaxation or tension. The music therapist will also demonstrate how to enter these effects into their daily music listening journal, which will be completed after each listening session.

Participants will be instructed to maintain their usual activities each day, except we will ask them to select a time of day, a comfortable and distraction free environment, and an apparatus for regular music listening (earbuds, headphones, speakers). Participants will listen mindfully to randomized selections from the playlist that meets their needs that day (i.e., energizing or relaxing). Participants will listen to their music selections on shuffle for 30 minutes per day for 8 weeks using the strategies provided by the music therapist. The target listening duration is 30 minutes as it is a common target for time spent on task before taking a break. Participants will complete their daily journal entry immediately after music listening.

The music therapist will make a weekly telephone call to each participant in the experimental arm. The telephone call will last ~30 minutes. During this telephone call, the music therapist will update the music playlists for the following week based on participant feedback. The music therapist will also inquire about the participant's daily music listening journals and help them submit their listening logs.

Active Control Arm (Audiobook Listening):

The active control group will follow the same protocol as the experimental (MBI) group, but instead of music, participants will listen to an audiobook of their choice for 30 minutes daily over 8 weeks. A trained speech-language pathologist, rather than a music therapist, will curate the audiobook playlist, provide listening strategies, guide participants on how to complete the listening session and journal entries, and conduct the weekly 30-minute phone calls. By standardizing listening duration and therapist interactions across both groups, any attention changes unique to the experimental group can be attributed to the effects of music, rather than general auditory input or human interaction.

No-Contact Control Arm (No Music or Audiobook Listening):

The no-contact control arm is designed to demonstrate that any behavioral changes observed in the experimental (MBI) arm are due to the intervention itself, rather than spontaneous recovery processes. While PWA did not achieve full recovery through spontaneous processes, they may still experience improvements over time that occur independently of therapeutic interventions. As such, participants in the no-contact control arm will be instructed to maintain their usual activities without any additional listening tasks. They will also not engage in weekly interactions with a therapist. The use of a no-contact control arm allows us to determine whether any changes observed in the experimental arm exceed those that might naturally occur without participation in the intervention.

Assessment Protocol: All participants will complete assessments of attention, language, and quality of life, at three timepoints: pre-intervention (T1), post-intervention (T2), and at the 8-week maintenance follow-up (T3). Participants will also answer questions about lifestyle factors such as regular caffeine intake, sleep patterns, medications, musical preferences, listening habits, and exercise routines that may impact the outcomes. The following assessments will be administered.

Attention Network Test (ANT): Attention will be measured using the ANT, which is a cued-flanker task developed to simultaneously measure alerting, one's readiness to perceive information; orienting, the ability to shift attention in response to a stimulus' properties; and executive control, the ability to focus on relevant information while simultaneously inhibiting irrelevant or distracting information. The ANT takes 10 minutes to complete and will be administered using Gorilla Experiment Builder. The PI's lab has extensive experience administering the ANT to PWA.

Each trial begins with a fixation cross displayed for a jittered duration of 2400-3600 ms. After the fixation cross offset, a visual cue appears for 100 ms. Cue conditions include: (1) spatial orienting cue (a single asterisk above or below the fixation cross), (2) double alerting cue (asterisks both above and below the fixation cross), (3) neutral orienting cue (a single asterisk in the center), and (4) neutral alerting cue (the fixation cross remains, i.e., no cueing is provided). After the cue offset, the fixation cross reappears for 400 ms, followed by the flanker task, which consists of five arrows that appear above or below the fixation cross. Participants indicate the direction of the center arrow via button press. Congruent trials have flanking arrows pointing in the same direction as the center arrow; incongruent trials have them pointing in the opposite direction; in neutral trials, dashed lines flank the center arrow. Participants are instructed to respond quickly and accurately. Participants complete 156 randomized trials, equally representing all cue types and flanker conditions. Verbal and written instructions, stimulus examples, and 10 practice trials precede the start of the task.

Extended Barcelona Music Reward Questionnaire (BMRQ) assesses participants' sensitivity to musical reward in six domains: Musical Seeking, Emotion Evocation, Mood Regulation, Social Reward, Sensory-Motor, and Absorption. Participants rate their agreement with 24 statements (4 per domain) using a 5-point Likert scale.

Goldsmiths Music Sophistication Index (GoldMSI) evaluates participant's ability to engage with music in an effective and flexible manner across 6 domains: Active Musical Involvement, Perceptual Listening Skills, Musical Training, Singing Abilities, Emotional Responses to Music, and Overall Musical Sophistication. PWA rate their agreement with 31 statements on a 7-point Likert scale and answer 8 forced-choice questions.

Language Production skills will be measured via a 5-minute monologue where PWA will talk about a topic(s) of their choosing from a provided list. Each sample will be videotaped, orthographically transcribed using CLAN, and coded for semantic (Word Finding Behavior Analysis; WFBA68) and syntactic production abilities (Quantitative Production Analysis; QPA69). For semantics (WFBA), we will mark paraphasias, neologisms, vague language, time fillers, and delays to calculate the percentage of word finding errors in the sample (%TWFB); %TWFB is a composite score that will be entered into the analyses. For syntax (QPA), we will code the sample for omitted words and sentence complexity (active, passive, etc.) and extract the proportion of well-formed sentences and complex sentences produced, which will be summed to produce a composite score that can be entered into the analyses.

Language Comprehension will be assessed using a computerized sentence-picture matching task. An auditory sentence will be presented binaurally at 60 decibels using headphones. Participants will simultaneously see two pictures (one target, one foil) and determine which picture matches the sentence as quickly (reaction time) and accurately as possible via a keyboard button press. Participants will complete 60 trials: 30 trials have a simple subject-verb-object sentence structure, and 30 trials have a complex subject-object-verb sentence structure. Trial presentation is randomized per participant. Verbal and written instructions, examples of all stimuli, and 5 practice trials will precede the start of the task. The dependent variables from this task are accuracy (proportion of correct responses) and mean reaction time across all sentences.

Quality of Life in Neurological Disorders (Neuro-QOL): Participants will complete select subtests from the Neuro-QOL, including the communication, participation in social roles and activities, anxiety, depression, and cognitive function subtests. PWA rate their agreement with items on a 5-point Likert scale. There are 8-9 items per subtest. Subtest scores will be summed and entered into the analyses.

ELIGIBILITY:
Inclusion Criteria:

Adults at least 18 years of age Individuals who have had a stroke and are at least 6 month post stroke Individuals are able to answer 4 questions to determine ability to consent (What is your name, what is the day/date, where are you , and why are we having this conversation).

Have normal or corrected to normal hearing Have normal or corrected to normal vision Have no issues with color blindness Individuals who have at least mild aphasia on the Western Aphasia Battery Revised Speaks American English

Exclusion Criteria:

Individuals who meet the inclusion criteria, but are unwilling to travel to the ABC Lab at Purdue University for in person testing and do not have a laptop or desktop with a web camera that they could participate online with, will be excluded.

Individuals who have had a dementia diagnosis or attention disorder pre stroke will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in attention from T1 to T2 and T3 | From T1 to T2 (11 weeks for the experimental and active control arms, 9 weeks for the no-contact arm) and to T3 (8 weeks after T2)
  Attention will be measured in each group through the Visual Attention Network Task. Changes in attention will be calculated between timepoint 1 (T1), timepoint 2 (T2) and timepoint 3 (T3).
Change in language from T1 to T2 and T3 | From T1 to T2 (11 weeks for the experimental and active control arms, 9 weeks for the no-contact arm) and to T3 (8 weeks after T2)
  Language will be measured through a sentence-picture matching task and language production task. Changes in language will be calculated between timepoint 1 (T1), timepoint 2 (T2) and timepoint 3 (T3).
Changes in quality of life from T1 to T2 and T3 | From T1 to T2 (11 weeks for the experimental and active control arms, 9 weeks for the no-contact arm) and to T3 (8 weeks after T2)
  Quality of life will be measured through the Quality of Life in Neurological Disorders measure. Changes in quality of life will be calculated between timepoint 1 (T1), timepoint 2 (T2) and timepoint 3 (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Arianna N LaCroix, PhD, Principal Investigator — Purdue University Speech, Language, and Hearing Science

IPD SHARING:
Plan to Share IPD: Yes
This project will generate behavioral data from one standardized language test, one 5 minute monologue, one experimental task of attention, one experimental task measuring language comprehension, one questionnaire regarding quality of life, and two questionnaires that assess participants' engagement and types of rewards experienced from music. All measures will be collected from all study participants pre- and post-intervention, and eight-weeks after the intervention concludes. The behavioral data will include verbal and written responses from the standardized tests and questionnaires, and reaction time and accuracy data from the experimental tasks. The standardized test and monologue will be videotaped. All de-identified data will be shared. We will not share the videotapes of the monologues as this information is identifiable.

REFERENCES:
- [Background] Varkanitsa M, Godecke E, Kiran S. How Much Attention Do We Pay to Attention Deficits in Poststroke Aphasia? Stroke. 2023 Jan;54(1):55-66. doi: 10.1161/STROKEAHA.122.037936. Epub 2022 Dec 21. PMID 36542078
- [Background] Dovorany N, Brannick S, Johnson N, Ratiu I, LaCroix AN. Happy and sad music acutely modulate different types of attention in older adults. Front Psychol. 2023 Jan 26;14:1029773. doi: 10.3389/fpsyg.2023.1029773. eCollection 2023. PMID 36777231